CLINICAL TRIAL: NCT05294731
Title: A Phase 1/2, Open-Label, Dose-Escalation and Expansion Study of the Bruton Tyrosine Kinase-Targeted Protein-Degrader BGB-16673 in Chinese Patients With B-Cell Malignancies
Brief Title: Treatment of Chinese Participants With B-Cell Malignancies With BGB-16673, a Bruton Tyrosine Kinase-Targeted Protein-Degrader
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-102; CTR20220399 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-02-22; First posted 2022-03-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: B-cell Malignancy; Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Waldenström Macroglobulinemia; Marginal Zone Lymphoma; Follicular Lymphoma; DLBCL Unclassifiable; Richter's Transformation
Keywords: B-cell Malignancy; MZL; FL; DLBCL; Richter's Transformation; CDAC; BTK; degrader; BGB-16673
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1a Monotherapy Dose Escalation (Experimental): BGB-16673 will be orally administered.
  Interventions: Drug: BGB-16673
- Phase 1b Monotherapy Safety Expansion (Experimental): BGB-16673 will be orally administered.
  Interventions: Drug: BGB-16673
- Phase 2 Monotherapy Dose Expansion (Experimental): BGB-16673 will be administered at the recommended Phase 2 dose (RP2D) that was identified in Part 1.
  Interventions: Drug: BGB-16673

INTERVENTIONS:
Drug: BGB-16673 — Orally administered

SUMMARY:
This study aims to explore the recommended phase 2 dose and evaluate the safety, tolerability and preliminary antitumor activity of BGB-16673 monotherapy at the recommended Phase 2 dose for the selected B-cell malignancy expansion cohorts

ELIGIBILITY:
Key Inclusion Criteria

1. Provision of signed and dated written informed consent prior to any study
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
3. Adequate organ function of coagulation function, liver function, renal function and pancreatic function and measure disease per disease-specific response criteria
4. Phase 1: Confirmed diagnosis of R/R Marginal Zone Lymphoma (MZL), Follicular Lymphoma (grade 1-3a), Waldenström Macroglobulinemia (WM), non-germinal center B-cell (non-GCB) diffuse large B-cell lymphoma (DLBCL), Richter's transformation to DLBCL, MCL, or CLL/SLL
5. Phase 2: Confirmed diagnosis of MCL, or CLL/SLL
6. Highly effective method of birth control during study treatment period, and for at least 90 days after the last dose of the study drug

Key Exclusion Criteria

1. Prior malignancy (other than the disease under study) within the past 2 years, except for curatively treated basal or squamous skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score ≤ 6 prostate cancer
2. Require ongoing systemic treatment for any other malignancy or systemic corticosteroid treatment
3. Receiving treatment with a strong CYP3A inhibitor or inducer ≤ 14 days before the first dose of BGB-16673, or proton-pump inhibitors ≤ 5 days before the first dose of BGB-16673.
4. Current or history of central nervous involvement
5. Prior autologous stem cell transplant unless ≥ 3 months after transplant, prior chimeric cell therapy unless ≥ 6 months after cell infusion, prior allogeneic stem cell transplant ≤ 6 months before the first dose of the study drug

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From first dose of the study drug(s) to 30 days after the last dose or before initiation of a new anticancer therapy, whichever occurs first (up to approximately 3 years)
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE 5.0), including AEs that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1: Recommended Phase 2 dose (RP2D) of BGB-16673 | From the date of first dose of study drugs until RP2D is determined (up to approximately 37 weeks)
  As determined by the sponsor based on the Safety Monitoring Committee's recommendation considering totality of the available clinical safety, clinical efficacy, pharmacokinetics, and pharmacodynamics data.
Phase 1a: Maximum tolerated dose (MTD) of BGB-16673 | From the date of first dose of study drugs until RP2D is determined (up to approximately 37 weeks)
  The highest dose evaluated as recommended by the Bayesian Optimal Interval Design with Informative Prior (iBOIN) design or the maximum assessed dose (MAD).
Phase 2: Overall Response Rate (ORR) in participants with Relapsed/Refractory (R/R) Mantle Cell Lymphoma (MCL) | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial response or better according to the Independent Review Committee (IRC) assessment and as determined by Lugano criteria.
Phase 2: ORR in participants with R/R Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial response or better as assessed by the IRC and determined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for CLL and by Lugano criteria for SLL

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Time to reach maximum observed plasma concentration (Tmax) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Minimum observed plasma concentration (Cmin) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Apparent terminal elimination half-life (t1/2) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Area under the plasma-concentration curve (AUC) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Apparent oral clearance (CL/F) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Apparent volume of distribution (Vz/F) After a Single Dose of BGB-16673 | Phase 1a: Week 1 Day 1 pre-dose up to 72 hours post-dose; Phase 1b: Week 1 Day 1 pre-dose and up to 6 hours post-dose; Phase 2: Week 1 Day 1 pre-dose and up to 8 hours post-dose
Maximum observed steady state plasma concentration (Css,max) of of BGB-16673 | Phase 1a and Phase 2: Week 5 Day 1 pre-dose and up to 8 hours post-dose; Phase 1b: Week 5 Day 1 pre-dose and up to 6 hours post-dose
Time to reach maximum observed steady state plasma concentration (Tss,max) of BGB-16673 | Phase 1a and Phase 2: Week 5 Day 1 pre-dose and up to 8 hours post-dose; Phase 1b: Week 5 Day 1 pre-dose and up to 6 hours post-dose
Minimum observed steady state plasma concentration (Css,min) of BGB-16673 | Phase 1a and Phase 2: Week 5 Day 1 pre-dose and up to 8 hours post-dose; Phase 1b: Week 5 Day 1 pre-dose and up to 6 hours post-dose
Steady state area under the plasma concentration-time curve (AUC) of BGB-16673 | Phase 1a and Phase 2: Week 5 Day 1 pre-dose and up to 8 hours post-dose; Phase 1b: Week 5 Day 1 pre-dose and up to 6 hours post-dose
Accumulation ratios of Cmax and AUC of BGB-16673 | Phase 1a: Day 1 pre-dose up to 72 hours post-dose, Week 5 pre-dose up to 8 hours post-dose; Phase 1b: Week 1 and Week 5 pre-dose up to 6 hours post-dose; Phase 2: Week 1 and Week 5 pre-dose up to 8 hours post-dose
Bruton's tyrosine kinase (BTK) protein degradation in peripheral blood after BGB-16673 monotherapy | Phase 1a: Day 1 pre-dose up to 72 hours post-dose, Week 5 pre-dose and 8 hours post-dose, Week 9 pre-dose; Phase 1b: Week 1 and Week 5 pre-dose and 6 hours post-dose, Week 9 pre-dose; Phase 2: Week 1, Week 5, Week 9 pre-dose
Phase 1: Overall Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial or complete response, as assessed by the investigator using International Workshop on Chronic Lymphocytic Leukemia (iwCLL), Owen, and Lugano criteria.
Phase 1: Major Response Rate (MRR) in participants with Waldenstrom macroglobulinemia (WM) | Up to approximately 3 years
  MRR is defined as the percentage of participants who achieved complete response (CR), very good partial response (VGPR), and partial response (PR), as assessed by investigators for participants with WM only.
Phase 2: Number of participants with AEs and SAEs | From first dose of the study drug(s) to 30 days after the last dose or before initiation of a new anticancer therapy, whichever occurs first (up to approximately 3 years)
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE 5.0).
Phase 2: ORR in participants with R/R MCL as assessed by investigators | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial response or better according to investigators and as determined by Lugano criteria.
Phase 2: Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first as determined by IRC and by investigators.
Phase 2: Time to Response (TTR) | Up to approximately 3 years
  TTR is defined as the time from study treatment start to date of the earliest qualifying response (partial response or better) as determined by IRC and by investigators.
Phase 2: Progression Free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as determined by IRC and by investigators.
Phase 2: Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from first study drug administration to the date of death due to any cause.
Phase 2: Best Overall Response (BOR) of Partial Response with Lymphocytosis (PR-L) in Participants with R/R CLL/SLL | Up to approximately 3 years
  BOR of PR-L or better as determined by IRC and by investigators per iwCLL criteria for CLL and per Lugano criteria for SLL
Phase 2: Change from baseline in National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Cancer Symptom Index-18 (NFLymSI-18) Disease-related Symptom Physical and Treatment Side Effect Subscales in participants with R/R MCL | Baseline and Day 1 of weeks 5, 13, 25, and 37
  The NFLymSI-18 questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and is divided into a total score. A mixed model for repeated measures (MMRM) will be used to estimate the mean change from baseline for NFlymSI-18 subscales of Disease-Related Symptoms Physical (DRSP), and "treatment side effects" (TSE).
Phase 2: ORR assessed by the Investigator in participants with R/R CLL/SLL | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial response or better as determined by investigators per iwCLL criteria for CLL and Lugano criteria for SLL.
Phase 2: Mean change from baseline for the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu ) questionnaire Physical Well-being and Functional Well-being Subscales for participants with R/R CLL/SLL | Baseline and Day 1 of weeks 5, 13, 25, and 37
  FACT-Leu is a 44-item patient reported outcome questionnaire with five subscales used to measure health-related quality of life (HRQoL) in leukemia patients. Each question is scored from 0 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (29):
- China (29):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chao Yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Army Medical University (Xinqiao Hospital), Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine Branch Yuhang, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/